CLINICAL TRIAL: NCT03205150
Title: A 12-week Randomized, Patient and Investigator Blinded, Placebo-controlled, Parallel Group Study to Investigate the Efficacy of LIK066 in Obese Patients With Non-alcoholic Steatohepatitis (NASH)
Brief Title: Effect of LIK066 on Reduction of Fatty Content in Livers of Obese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIK066X2204; 2017-002046-71 (EudraCT Number)
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Results first posted 2021-01-06 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Obese Patients With Non-alcoholic Steatohepatitis (NASH)
Keywords: non-alcoholic steatohepatitis; NASH; Obese; Type 2 diabetes mellitus; non-alcoholic fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Diabetes Mellitus, Type 2 | interventions — licogliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LIK066 30 mg (Experimental): Film coated tablet of LIK066 30 mg was mostly administered once daily before lunch, except on Day 56 when it was administered before breakfast and in fasted state on Day 84.
  Interventions: Drug: LIK066
- LIK066 150 mg (Experimental): Film coated tablet of LIK066 150 mg was mostly administered once daily before lunch, except on Day 56 when it was administered before breakfast and in fasted state on Day 84
  Interventions: Drug: LIK066
- Placebo (Experimental): LIK066 0 mg film-coated tablet(Placebo matching tablets) was mostly administered once daily before lunch, except on Day 56 when it was administered before breakfast and in fasted state on Day 84.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIK066 — Film coated tablet of LIK066 either 30mg or 150 mg was mostly administered once daily before lunch, except on Day 56 when it was administered before breakfast and in fasted state on Day 84
  Arms: LIK066 150 mg; LIK066 30 mg
Drug: Placebo — LIK066 0 mg film-coated tablet(Placebo matching tablets) was mostly administered once daily before lunch, except on Day 56 when it was administered before breakfast and in fasted state on Day 84.
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the effects of LIK066 on a variety of metabolic and inflammation biomarkers in patients with non-alcoholic steatohepatitis (NASH)

DETAILED DESCRIPTION:
This was a a non-confirmatory, multicenter, patient and investigator blinded, randomized, placebo-controlled, parallel group study in patients with non-alcoholic steatohepatitis (NASH).

The study consisted of a 28 day screening period (Day -44 to Day -16), a baseline period of 14 days (Day -15 to Day -1), a treatment period of 12 weeks (Day 1 to Day 84), and a study completion evaluation approximately 28 days after the last drug administration. The patients were advised to maintain their recommended diet during the study.

Patients who met the inclusion/exclusion criteria at screening went to the study site for baseline assessments. All baseline safety evaluation results were available prior to the first dosing.

The study started by enrolling patients into the 150 mg and placebo arms with a randomization ratio of 2:1. After the enrollment of the first 33 patients, the 30 mg arm was added to the study and the randomization ratio changed to a 2:4:1 ratio (150 mg: 30 mg: placebo) to maintain the 2:2:1 ratio across the three groups (150 mg: 30 mg: placebo) at study completion.

ELIGIBILITY:
Inclusion Criteria:

EITHER

-Histologic confirmed NASH based on liver biopsy obtained 2 years or less before randomization with a fibrosis level of F1, F2 or F3 in the absence of a histological diagnosis of alternative chronic liver disease AND ALT greater than or equal to 50 IU/L (males) or greater than or equal to 35 IU/L (females) at screening.

OR

Phenotypic diagnosis of NASH based on presence of ALL three of the following at screening:

* ALT greater than or equal to 50IU/L (males) or greater than or equal to 35 IU/L (females) AND
* BMI greater than or equal to 27 kg/m^2 (in patients with a self-identified race other than Asian) or greater than or equal to 23 kg/m^2 (in patients with a self identified Asian race) AND
* Diagnosis of Type 2 diabetes mellitus by HbA1c: greater than or equal to 6.5 % and less than or equal to 10%
* Patients must weigh no more than 150 kg (330 lbs) to participate in the study.
* Male and female patients 18 years or older at the time of screening visit.

Exclusion Criteria:

* History or presence of other concomitant liver diseases
* History or current diagnosis of ECG abnormalities
* Use of GLP-1 agonists, SGLT2 inhibitors, TZDs, FXR agonists and any pharmacologically active weight loss drugs within 6 weeks of screening and until end of study
* Patients with contraindications to MRI imaging
* Current or history of significant alcohol consumption
* Clinical evidence of hepatic decompensation or severe liver impairment
* Women of child bearing potential (unless on basic contraception methods)
* Presence of liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (4):
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Live Oak, Texas
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Novartis Investigative Site, Montreal, Quebec, Canada
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Novartis Investigative Site, Leiden, Netherlands
- Novartis Investigative Site, Saint Petersburg, Russia
- Taiwan (2):
  - Novartis Investigative Site, Chiayi City
  - Novartis Investigative Site, Tainan
- Novartis Investigative Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Harrison SA, Manghi FP, Smith WB, Alpenidze D, Aizenberg D, Klarenbeek N, Chen CY, Zuckerman E, Ravussin E, Charatcharoenwitthaya P, Cheng PN, Katchman H, Klein S, Ben-Ari Z, Mendonza AE, Zhang Y, Martic M, Ma S, Kao S, Tanner S, Pachori A, Badman MK, He Y, Ukomadu C, Sicard E. Licogliflozin for nonalcoholic steatohepatitis: a randomized, double-blind, placebo-controlled, phase 2a study. Nat Med. 2022 Jul;28(7):1432-1438. doi: 10.1038/s41591-022-01861-9. Epub 2022 Jun 20. PMID 35725922
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 107 participants were enrolled in 15 centers across 8 countries: Argentina (2), Canada (1), Israel (3), Netherlands (1), Russia federation (1), Taiwan (2), Thailand (1), United States (4).
Pre-assignment Details: Participants were randomized in 2:2:1 ratio to the 3 groups: LIK066 150 mg, LIK066 30 mg and placebo.
Period: Overall Study
Arm/Group | LIK066 30 mg | LIK066 150 mg | Placebo
Started (Participants randomized) | 43 | 43 | 21
Safety Analysis Set | 43 | 43 | 21
Pharmacokinetics (PK) Analysis Set | 42 (all patients with valid PK measurements) | 36 (all patients with valid PK measurements) | 0 (Placebo patients were excluded from the PK analyses)
Pharmacodynamics (PD) Analysis Set | 43 (all patients with available PD data and no protocol deviations) | 41 (all patients with available PD data and no protocol deviations) | 21 (all patients with available PD data and no protocol deviations)
Completed | 41 | 36 | 19
Not Completed | 2 | 7 | 2
Not completed — Protocol deviation | 1 | 3 | 0
Not completed — Patient/guardian decision | 0 | 3 | 0
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LIK066 30 mg | LIK066 150 mg | Total
Number analyzed (Participants) | 21 | 43 | 43 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (11.16) | 53.1 (12.57) | 49.5 (11.10) | 50.7 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 25 | 22 | 59
  Male | 9 | 18 | 21 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 34 | 35 | 86
  Asian | 3 | 8 | 4 | 15
  Black or African American | 1 | 1 | 3 | 5
  Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alanine Aminotransferase (ALT) at Week 12
Description: Alanine aminotransferase (ALT) is an enzyme found primarily in the liver. ALT is increased with liver damage. In this study, the blood levels of ALT was used to detect liver injury. Baseline is defined as the mean of measurements taken at the Screening and Baseline visits.
Time Frame: Baseline, Week 12
Population: Pharmacodynamics (PD) analysis set: included all participants with available PD data, who received any study drug and had valid measurements for the outcome measure
Measure: Mean (Standard Error); unit: Units per Liter (U/L)
Arm/Group | LIK066 30 mg | LIK066 150 mg | Placebo
Number analyzed (Participants) | 40 | 34 | 20
Units per Liter (U/L) | -22.06 (4.16) | -30.41 (4.52) | -8.77 (5.99)
Statistical Analysis 1: Comparison: LIK066 30 mg vs Placebo; Test type: Superiority; p = 0.075, ANCOVA; Mean Difference (Net) = -13.29, 80% CI 2-sided [-22.80 to -3.78], Standard Error of Mean 7.35
Statistical Analysis 2: Comparison: LIK066 150 mg vs Placebo; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Net) = -21.64, 80% CI 2-sided [-31.33 to -11.94], Standard Error of Mean 7.49
Statistical Analysis 3: Comparison: LIK066 30 mg vs LIK066 150 mg; Test type: Superiority; p = 0.178, ANCOVA; Mean Difference (Net) = 8.35, 80% CI 2-sided [0.41 to 16.29], Standard Error of Mean 6.14

2. Secondary Outcome: Change From Baseline in Percent Liver Fat at Week 12
Description: Percent (%) Liver fat was measured by Magnetic Resonance Imaging Proton Density Liver Fat Fraction(MRIPDFF). Patients underwent magnetic resonance imaging twice during the course of the study ( baseline and end of treatment) to quantitate liver fat.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage of Liver Fat
Arm/Group | LIK066 30 mg | LIK066 150 mg | Placebo
Number analyzed (Participants) | 39 | 33 | 19
Percentage of Liver Fat | -4.40 (0.81) | -6.92 (0.87) | -2.67 (1.17)
Statistical Analysis 1: Comparison: LIK066 30 mg vs Placebo; Test type: Superiority; p = 0.235, ANCOVA; Mean Difference (Net) = -1.73, 80% CI 2-sided [-3.60 to 0.14], Standard Error of Mean 1.45
Statistical Analysis 2: Comparison: LIK066 150 mg vs Placebo; Test type: Superiority; p = 0.004, ANCOVA; Mean Difference (Net) = -4.26, 80% CI 2-sided [-6.14 to -2.37], Standard Error of Mean 1.46
Statistical Analysis 3: Comparison: LIK066 30 mg vs LIK066 150 mg; Test type: Superiority; p = 0.037, ANCOVA; Mean Difference (Net) = 2.52, 80% CI 2-sided [0.98 to 4.07], Standard Error of Mean 1.19

3. Secondary Outcome: Percent Change From Baseline in Total Body Weight at Week 12
Description: Body weight (to the nearest 0.1 kilogram [kg] was measured on a calibrated scale. The measurement was performed with the study subject in underwear and without shoes; or while wearing minimal indoor clothing.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | LIK066 30 mg | LIK066 150 mg | Placebo
Number analyzed (Participants) | 40 | 34 | 19
percentage change | -3.48 (0.47) | -4.51 (0.52) | -0.33 (0.68)
Statistical Analysis 1: Comparison: LIK066 30 mg vs Placebo; Test type: Superiority; p < .001, ANCOVA; Mean Difference (Net) = -3.15, 80% CI 2-sided [-4.22 to -2.08], Standard Error of Mean 0.83
Statistical Analysis 2: Comparison: LIK066 150 mg vs Placebo; Test type: Superiority; p < .001, ANCOVA; Mean Difference (Net) = -4.18, 80% CI 2-sided [-5.28 to -3.08], Standard Error of Mean 0.85
Statistical Analysis 3: Comparison: LIK066 30 mg vs LIK066 150 mg; Test type: Superiority; p = 0.148, ANCOVA; Mean Difference (Net) = 1.03, 80% CI 2-sided [0.12 to 1.94], Standard Error of Mean 0.71

4. Secondary Outcome: Change From Baseline in Non-invasive Markers of Hepatic Fibrosis: Enhanced Liver Fibrosis Test (ELF) Score at Week 12
Description: The markers of fibrosis assessed in this test comprised hyaluronic acid (HA), tissue inhibitor of metalloproteinase (TIMP1) and procollagen III N-terminal peptide (PIIINP); these are components of the extracellular matrix and basement sinusoidal membrane of the liver and are elevated during fibrogenesis as a result of activation of the hepatic stellate cell. The ELF test is a composite score: < 7.7: no to mild fibrosis; ≥ 7.7 - < 9.8: Moderate fibrosis; ≥ 9.8 - < 11.3: Severe fibrosis; ≥ 11.3: Cirrhosis. A negative change from Baseline indicates decreased fibrosis.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | LIK066 30 mg | LIK066 150 mg | Placebo
Number analyzed (Participants) | 40 | 34 | 21
scores on a scale | -0.2 (0.65) | -0.1 (0.61) | 0.1 (0.37)

5. Secondary Outcome: Change From Baseline in the Concentration of Hyaluronic Acid at Week 12.
Description: Hyaluronic Acid is a non-invasive marker of liver fibrosis. It was accessed by Enhanced liver fibrosis Test (ELF).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | LIK066 30 mg | LIK066 150 mg | Placebo
Number analyzed (Participants) | 40 | 34 | 21
ug/L | -3.4 (75.38) | 0.4 (30.56) | 4.7 (21.73)

6. Secondary Outcome: Change From Baseline in the Concentration of Procollagen Type Iii N-Terminal Peptide (PIIINP) at Week 12.
Description: PIIINP is a non-invasive marker of liver fibrosis. It was accessed by Enhanced liver fibrosis Test (ELF).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | LIK066 30 mg | LIK066 150 mg | Placebo
Number analyzed (Participants) | 40 | 34 | 20
ug/L | -1.7 (2.73) | -1.2 (3.66) | 0.3 (1.88)

7. Secondary Outcome: Change From Baseline in the Concentration of Tissue Inhibitor Of Metalloproteinase 1 (TIMP-1) at Week 12.
Description: TIMP-1 is a non-invasive marker of liver fibrosis. It was accessed by Enhanced liver fibrosis Test (ELF).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | LIK066 30 mg | LIK066 150 mg | Placebo
Number analyzed (Participants) | 40 | 34 | 20
ug/L | -3.0 (38.98) | -10.9 (38.21) | 10.3 (25.73)

8. Secondary Outcome: Pharmacokinetics of LIK066: Observed Maximum Plasma Concentration (Cmax) Following Drug Administration
Description: Cmax is the observed maximum plasma concentration following drug administration (ng/mL)
Time Frame: Day 56 (pre-dose and 1, 2, 4 and 6 hours post-dose)
Population: Pharmacokinetics (PK) analysis set consisted of LIK066 treated patients. Placebo patients were excluded from the PK analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LIK066 30 mg | LIK066 150 mg
Number analyzed (Participants) | 38 | 32
ng/mL | 405 (109) | 1810 (729)

9. Secondary Outcome: Pharmacokinetics of LIK066: Observed Maximum Time Duration of Maximum Concentration (Tmax) Following Drug Administration
Description: Tmax is the time to reach the maximum concentration after drug administration (hour). The time points presented are the actual and not the planned time points.
Time Frame: Day 56 (pre-dose and 1, 2, 4 and 6 hours post-dose)
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | LIK066 30 mg | LIK066 150 mg
Number analyzed (Participants) | 38 | 32
hours | 1.00 [0.500 to 6.00] | 1.51 [0.567 to 6.00]

10. Secondary Outcome: Pharmacokinetics of LIK066: Observed Area Under the Curve up to the Last Measurable Concentration (AUClast) Following Drug Administration
Description: AUClast is the area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (hour*ng/mL)
Time Frame: Day 56 (pre-dose and 1, 2, 4 and 6 hours post-dose)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | LIK066 30 mg | LIK066 150 mg
Number analyzed (Participants) | 38 | 32
hour*ng/mL | 1280 (413) | 5770 (1680)

11. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) at Week 12
Description: Aspartate aminotransferase (AST) is an enzyme found in many cells of the body specifically those of the liver, heart and skeletal muscle. In healthy individuals, levels of AST in the blood are low. When liver or muscle cells are injured, they release AST into the blood. In this study, the blood levels of AST was used to detect liver injury. Baseline is defined as the mean of measurements taken at the Screening and Baseline visits.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units per liter (U/L)
Arm/Group | LIK066 30 mg | LIK066 150 mg | Placebo
Number analyzed (Participants) | 40 | 34 | 20
Units per liter (U/L) | -13.45 (2.46) | -17.01 (2.68) | -2.30 (3.54)
Statistical Analysis 1: Comparison: LIK066 30 mg vs Placebo; Test type: Superiority; p = 0.013, ANCOVA; Mean Difference (Net) = -11.15, 80% CI 2-sided [-16.79 to -5.50], Standard Error of Mean 4.36
Statistical Analysis 2: Comparison: LIK066 150 mg vs Placebo; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Net) = -14.71, 80% CI 2-sided [-20.43 to -8.98], Standard Error of Mean 4.43
Statistical Analysis 3: Comparison: LIK066 30 mg vs LIK066 150 mg; Test type: Superiority; p = 0.332, ANCOVA; Mean Difference (Net) = 3.56, 80% CI 2-sided [-1.15 to 8.28], Standard Error of Mean 3.65

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of study treatment until the end of study treatment i.e. Day 84 plus 28 days recovery and follow-up period.
Description: Any signs or symptoms that occured from the first dose of study treatment until the end of study treatment i.e. Day 84 plus 28 days recovery and follow-up period.
Groups:
- All Patients: All Patients
Arm/Group | LIK066 30 mg | LIK066 150 mg | Placebo | All Patients
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/21 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 1/21 | 1/107
Other Adverse Events (participants affected / at risk) | 31/43 | 36/43 | 18/21 | 85/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LIK066 30 mg (N=43) | LIK066 150 mg (N=43) | Placebo (N=21) | All Patients (N=107)
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LIK066 30 mg (N=43) | LIK066 150 mg (N=43) | Placebo (N=21) | All Patients (N=107)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 6 | 0 | 8
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 2 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 2 | 5
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 21 | 33 | 9 | 63
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Flatulence (Gastrointestinal disorders) | 2 | 8 | 2 | 12
Gastric dilatation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 3 | 3 | 10
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 5 | 2 | 2 | 9
Asthenia (General disorders) | 1 | 1 | 1 | 3
Chills (General disorders) | 0 | 0 | 1 | 1
Early satiety (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 2 | 3 | 0 | 5
Feeling hot (General disorders) | 0 | 0 | 1 | 1
Feeling jittery (General disorders) | 0 | 0 | 1 | 1
Hunger (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 2
Thirst (General disorders) | 0 | 1 | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 1
Furuncle (Infections and infestations) | 1 | 0 | 1 | 2
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1
Gingival abscess (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 4 | 0 | 0 | 4
Nasopharyngitis (Infections and infestations) | 0 | 3 | 1 | 4
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 4
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 3
Vaginal infection (Infections and infestations) | 0 | 2 | 0 | 2
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 1
Heart rate irregular (Investigations) | 0 | 1 | 0 | 1
Lymphocyte morphology abnormal (Investigations) | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Polydipsia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 4
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 4 | 3 | 7
Head discomfort (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 5 | 3 | 10
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 1
Ketonuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Microalbuminuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 1
Polyuria (Renal and urinary disorders) | 4 | 1 | 1 | 6
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Diastolic hypotension (Vascular disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT03205150/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT03205150/SAP_001.pdf